CLINICAL TRIAL: NCT03654170
Title: Metabolism and Pharmacokinetics of BI 425809 After Administration of BI 425809 (C-14) as Oral Solution in Healthy Male Volunteers
Brief Title: A Study in Healthy Men to Find Out How BI 425809 is Taken up and Handled by the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0016; 2018-001192-21 (EudraCT Number)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Carbon-14

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): BI 425809 mixed with [C14] BI 425809
  Interventions: Drug: BI 425809 mixed with [C-14] BI425809

INTERVENTIONS:
Drug: BI 425809 mixed with [C-14] BI425809 — Oral Solution
  Other Names: Iclepertin

SUMMARY:
This trial intends to investigate the basic pharmacokinetics of BI 425809 and [14C]- radioactivity, including mass balance, excretion pathways and metabolism following a single oral dose of 25 mg BI 425809 (C-14) given to healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 65 years (incl.)
* BMI of 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation
* Subjects who are sexually active must use, with their partner, highly effective contraception from the time of administration of trial medication until 4 months after administration of trial medication.
* Subjects are required to use condoms to prevent unintended exposure of the partner to the study drug via seminal fluid. Alternatively, true abstinence is acceptable when it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active but becomes active, with their partner, they must comply with the contraceptive requirements detailed above.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 139 mmHg, diastolic blood pressure outside the range of 45 to 89 mmHg, or pulse rate outside the range of 40 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Clinically significant gastrointestinal, hepatic, renal, respiratory (including but not limited to interstitial lung disease), cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation). Use of CYP3A4 inhibitors and inducers 1 week prior to administration of trial medication
* Participation in another trial where an investigational drug has been administered within 60 days prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 5 cigarettes or 1 cigars or 1 pipes per day)
* Inability to refrain from smoking on trial days
* Average intake of more than 24 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 ml of spirits)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within 4 days prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
feurine, 0-t2 (fraction of [14C]-radioactivity excreted in urine as percentage of the administered oral dose over the time interval from 0 to the last quantifiable time point) | Up to 7 weeks
fefaeces, 0-t2 (fraction of [14C]-radioactivity excreted in faeces as percentage of the administered oral dose over the time interval from 0 to the last quantifiable time point) | Up to 7 weeks

SECONDARY OUTCOMES:
Cmax (maximum measured concentration of the analyte) | Up to 7 weeks
AUC0-tz (area under the concentration-time curve of the analyte over the time interval from 0 to the last quantifiable time point) | Up to 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences Onderzoekscentrum Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. Studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. Studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement.

REFERENCES:
- [Derived] Burkard U, Desch M, Shatillo Y, Wunderlich G, Mack SR, Schlecker C, Teitelbaum AM, Liu P, Chan TS. The Absolute Bioavailability, Absorption, Distribution, Metabolism, and Excretion of BI 425809 Administered as an Oral Dose or an Oral Dose with an Intravenous Microtracer Dose of [14C]-BI 425809 in Healthy Males. Clin Drug Investig. 2022 Jan;42(1):87-99. doi: 10.1007/s40261-021-01111-9. Epub 2021 Dec 22. PMID 34936055